CLINICAL TRIAL: NCT03374683
Title: Go Play Outside! Effects of a Risk Reframing Tool on Mothers' Tolerance for and Parenting Practices Associated With Children's Risky Play - a Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of a Risk Reframing Tool to Change Mothers' Parenting Associated With Children's Risky Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Mariana Brussoni, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H15-03271
Record Dates: First submitted 2017-12-06; First posted 2017-12-15 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Risk Assessment; Parenting
Keywords: Risky play; Physical activity; Injury prevention; Outdoor play
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RR Digital Tool (Experimental): Participants in the RR digital tool were provided with a link to the web-based intervention (https://outsideplay.ca) to complete within one week.
  Interventions: Behavioral: RR Digital Tool
- RR In-Person Workshop (Active Comparator): Participants in the in-person workshop attended the 45-90 minute in-person workshop.
  Interventions: Behavioral: RR In-Person Workshop
- Position Statement on Active Outdoor Play (Sham Comparator): Participants in the control condition were provided with a web link to the Position Statement on Active Outdoor Play, which includes information on research and recommendations for action.
  Interventions: Behavioral: Position Statement on Active Outdoor Play

INTERVENTIONS:
Behavioral: RR Digital Tool — Participants proceed through three chapters in the tool: https://outsideplay.ca.
  Chapter 1: most important attributes they want for their child; their child's favourite play activities; their own childhood play activities; how their child's and their own play activities compare.
  Chapter 2: imagining themselves in three video segments where they must decide whether they allow their child to climb a tree, walk home from school, and use box cutters to build a fort. They reflect on their barriers and things that helped them let go.
  Chapter 3: revisiting the most important attributes they want for their child and whether there is anything they want to change, setting a realistic goal, outlining steps for attaining that goal, and setting start date.
  Arms: RR Digital Tool
Behavioral: RR In-Person Workshop — Participants engage in a facilitator guided discussion of the same tasks as the RR digital tool. Participants are taken through each task using PowerPoint slides that include the videos from the digital tool. The facilitator guide contains detailed guidance on discussion for each component and length of time to be dedicated to each slide. Participants are provided with a paper booklet to complete that mimics the online tasks.
  Arms: RR In-Person Workshop
Behavioral: Position Statement on Active Outdoor Play — The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety (ParticipACTION Canada, 2015; Tremblay et al., 2015).
  Arms: Position Statement on Active Outdoor Play

SUMMARY:
Children's risky play is associated with a variety of positive developmental, physical and mental health outcomes, including greater physical activity, self-confidence and risk management skills. Children's opportunities for risky play have eroded over time, limited by parents' fears and beliefs about risk, particularly among mothers. We have developed a digital and in-person workshop version of a tool to reframe parents' perceptions of risk. We examined whether the tool increased mothers' tolerance for risky play and influenced parenting behaviour change, in the short and long term, and whether these changes were greater than those in the control group.

We conducted a single-blind (researchers and outcome assessors) randomized controlled trial and recruited a total of 410 mothers of children aged 6-12 years. The risk reframing (RR) digital tool is designed for a one-time visit and includes three chapters of self-reflection and experiential learning tasks. The RR in-person tool is a 45-90 minute facilitated workshop in which participants were guided through discussions of the same tasks contained within the digital tool. The control condition consisted of reading the Position Statement on Active Outdoor Play.

Primary outcome was increased tolerance of risk in play, as measured by the Tolerance of Risk in Play Scale. Secondary outcome was self-reported attainment of a behaviour change goal that participants had set for themselves. We tested the hypothesis that there would be differences between the experimental and control groups with respect to tolerance of risk in play and goal attainment.

DETAILED DESCRIPTION:
The study used 3-group parallel randomized controlled trial design.

Participants were recruited through advertising on social media, distributing notices through our networks, snowball sampling, and posting notices in community centres. The aim was to obtain complete data on 375 participants. Interested participants completed a questionnaire in REDCap electronic data capture tool hosted at British Columbia Children's Hospital Research Institute to answer eligibility questions and provide informed consent. Enrolled participants received a link to the baseline questionnaire package to be completed in REDcap.

Once participants were deemed eligible for the study, they were allocated to one of the three conditions: 1) Control group; 2) RR digital tool; and 3) RR in-person workshop. Participants in Condition 1 were provided with a link to the Position Statement on Active Outdoor Play, which included information on research and recommendations for action. Participants in Condition 2 were provided with a link to the RR digital tool to complete at their leisure. Participants in Condition 3, were scheduled to attend the RR in-person workshop. The randomization schedule was generated beforehand in sealedenvelop.com using blocks of size 3, 6, and 9. The list was then transferred to REDCap.

Honoraria were paid at each time point as compensation for participation. Participants attending in-person RR workshops were provided with an additional honorarium to compensate them for any expenses incurred in attending, such as travel or childcare.

Participants had an equal likelihood of assignment to each condition (33%). The nature of the intervention did not permit participant blinding but they were informed of their allocated treatment after completing the baseline questionnaires. The in-person workshop facilitator could not be blinded to allocation as the other two arms did not have a facilitator. Likewise, research staff who coordinated in-person workshop schedules could not be blinded to the allocation of the in-person workshop. However, allocations were concealed to the researchers at participant assignment and data analysis.

Participants completed a questionnaire package at three time points: Baseline, 1-week post-intervention, and 3-months post-intervention. Survey data were collected and managed using REDCap.

The study hypotheses were:

1. Mothers completing the RR digital tool will have a significantly greater increase of tolerance for risk in play than mothers in the control condition.
2. Mothers completing the RR in-person workshop will have a significantly greater increase of tolerance for risk in play than mothers in the control condition.
3. A greater proportion of mothers completing the RR digital tool will attain their behaviour change goal, than mothers in the control condition.
4. A greater proportion of mothers completing the RR in-person workshop will attain their behaviour change goal than mothers in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Being a mother with primary custody of a child/children aged 6-12 years
* Residing in the Metro Vancouver Regional District
* Being able to speak, read and understand English

Exclusion Criteria:

* Being a father
* Not having a child between the ages of 6-12 years
* Not having primary custody of the child
* Not residing in Metro Vancouver Regional District
* Limited English skills

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant self-identifies as mother.
Enrollment: 451 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Brussoni, PhD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data set will be available from Dr. Brussoni upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting upon publication of the RCT results until five years after publication.
Access Criteria: Dr. Brussoni will review requests and share supporting information as indicated above with researchers and students doing similar research.

REFERENCES:
- [Background] Tremblay MS, Gray C, Babcock S, Barnes J, Bradstreet CC, Carr D, Chabot G, Choquette L, Chorney D, Collyer C, Herrington S, Janson K, Janssen I, Larouche R, Pickett W, Power M, Sandseter EB, Simon B, Brussoni M. Position Statement on Active Outdoor Play. Int J Environ Res Public Health. 2015 Jun 8;12(6):6475-505. doi: 10.3390/ijerph120606475. PMID 26062040
- [Background] Sandseter EB. Characteristics of risky play. J Adventure Educ Outdoor Learn. 2009;9(1):3-21. doi:10.1080/14729670802702762.
- [Background] Hill A, Bundy AC. Reliability and validity of a new instrument to measure tolerance of everyday risk for children. Child Care Health Dev. 2014 Jan;40(1):68-76. doi: 10.1111/j.1365-2214.2012.01414.x. Epub 2012 Jul 30. PMID 22846064
- [Background] ParticipACTION. The Biggest Risk Is Keeping Kids Indoors: ParticipACTION Report Card on Physical Activity for Children and Youth. Toronto, Ontario; 2015.
- [Background] Brussoni M, Ishikawa T, Han C, Pike I, Bundy A, Faulkner G, Masse LC. Go Play Outside! Effects of a risk-reframing tool on mothers' tolerance for, and parenting practices associated with, children's risky play: study protocol for a randomized controlled trial. Trials. 2018 Mar 7;19(1):173. doi: 10.1186/s13063-018-2552-4. PMID 29514699
- [Result] Brussoni M, Han CS, Lin Y, Jacob J, Pike I, Bundy A, Faulkner G, Gardy J, Fisher B, Masse L. A Web-Based and In-Person Risk Reframing Intervention to Influence Mothers' Tolerance for, and Parenting Practices Associated With, Children's Outdoor Risky Play: Randomized Controlled Trial. J Med Internet Res. 2021 Apr 27;23(4):e24861. doi: 10.2196/24861. PMID 33904820
- See also: Canadian Position Statement on Active Outdoor Play — https://www.outdoorplaycanada.ca/position-statement-on-active-outdoor-play/
- See also: Risk Reframing Digital Tool — https://outsideplay.ca/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertising on online forums and social media, distributing notices through our networks, snowball sampling and posting notices in community centers. Recruitments were active from December 2017 to May 2018 in the Metro Vancouver area.
Pre-assignment Details: Participants were randomized to a condition when they were deemed eligible. After being randomized, participants received the socio-demographic questionnaire and the intervention. A total of 451 participants who completed the socio-demographic questionnaire were included in the study.
Groups:
- Position Statement Active Outdoor Play: Position Statement Active Outdoor Play: The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety (ParticipACTION Canada, 2015; Tremblay et al., 2015).
- Risk Reframing (RR) Digital Tool: RR Digital Tool: Participants proceed through three chapters in the tool: https://outsideplay.ca. Chapter 1: most important attributes they want for their child; their child's favourite play activities; their own childhood play activities; how their child's and their own play activities compare.
  Chapter 2: imagining themselves in three video segments where they must decide whether they allow their child to climb a tree, walk home from school, and use box cutters to build a fort. They reflect on their barriers and things that helped them let go.
  Chapter 3: revisiting the most important attributes they want for their child and whether there is anything they want to change, setting a realistic goal, outlining steps for attaining that goal, and setting start date.
- RR In-Person Workshop: RR In-Person Workshop: Participants engage in a 2-hour facilitator guided discussion of the same tasks as the RR digital tool. Participants are taken through each task using PowerPoint slides that include the videos from the digital tool. The facilitator guide contains detailed guidance on discussion for each component and length of time to be dedicated to each slide. Participants are provided with a paper booklet to complete that mimics the online tasks.
Period: Overall Study
Arm/Group | Position Statement Active Outdoor Play | Risk Reframing (RR) Digital Tool | RR In-Person Workshop
Started | 148 | 150 | 153
1-week Post-intervention | 135 | 113 | 85
Completed | 123 | 105 | 84
Not Completed | 25 | 45 | 69

BASELINE CHARACTERISTICS:
Groups:
- Position Statement on Active Outdoor Play: Position Statement Active Outdoor Play: The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety (ParticipACTION Canada, 2015; Tremblay et al., 2015).
- Total: Total of all reporting groups
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool | RR In-Person Workshop | Total
Number analyzed (Participants) | 148 | 150 | 153 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (5.3) | 40.8 (5.5) | 39.6 (5.0) | 40.29 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 150 | 153 | 451
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Population groups: White | 101 | 112 | 117 | 330
  Population groups: Other | 47 | 38 | 36 | 121
Marital status [Count of Participants; unit: Participants]
  Married/Common-law | 118 | 125 | 131 | 374
  Other | 30 | 25 | 22 | 77
Education [Count of Participants; unit: Participants]
  < university / college | 36 | 36 | 33 | 105
  University / college | 66 | 80 | 72 | 218
  > university college | 46 | 32 | 46 | 124
  Missed data | 0 | 2 | 2 | 4
Employment [Count of Participants; unit: Participants]
  Employed for wages/self employed | 115 | 107 | 44 | 266
  Unemployed | 33 | 43 | 109 | 185
Home dwelling [Count of Participants; unit: Participants]
  Single-detached | 69 | 77 | 72 | 218
  Others | 79 | 73 | 81 | 233
Income [Count of Participants; unit: Participants]
  < $63,300 | 36 | 40 | 33 | 109
  $63,300-$103,299 | 49 | 40 | 50 | 139
  >=$103,300 | 52 | 54 | 55 | 161
  Prefer not to answer | 11 | 16 | 15 | 42
Exposure to risky play information [Count of Participants; unit: Participants] — Participants were asked in the socio-demographic questionnaire, if they had been exposed to any information on risky play in the context of children's outdoor play. This was to understand if participants had been primed or tainted by any previous knowledge or training on children's outdoor risky play before participating in our study. The question reads, 'In the last month, have you seen any information on risky play?', which can be answered 'yes' or 'no'.
  Participants
    No | 126 | 122 | 117 | 365
    Yes | 22 | 28 | 36 | 86
Child age [Mean (Standard Deviation); unit: years] | 8.4 (1.7) | 8.1 (1.7) | 8.0 (1.9) | 8.1 (1.8)
Child sex [Count of Participants; unit: Participants]
  Boy | 85 | 82 | 85 | 252
  Girl | 60 | 68 | 67 | 195
  Missing data | 3 | 0 | 1 | 4
Child's disability/chronic condition [Count of Participants; unit: Participants] — Participants were asked in the socio-demographic questionnaire, if their child had any disability or long-term health problem that could limit her/his normal physical outdoor risky play. This was to understand if participants' risk tolerance in children's play were influenced by their child's disability or long-term health conditions. The question reads, 'Does your child suffer from a disability or long-term health problem that limits her/his normal activities?', which can be answered 'yes' or 'no'.
  Participants
    No | 143 | 140 | 148 | 431
    Yes | 5 | 10 | 5 | 20
Outdoor time [Mean (Standard Deviation); unit: hours]
  Weekday | 3.0 (3.6) | 2.8 (3.2) | 2.6 (2.8) | 2.80 (3.20)
  Weekend | 2.7 (2.2) | 2.8 (2.0) | 2.9 (2.8) | 2.79 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tolerance of Risk in Play Scale (TRiPS)
Description: The primary outcome measure was increase in the total score on the Tolerance for Risk in Play Scale (TRiPS), a 31-item measure examining adults' tolerance of risk during children's play. This analysis was conducted using mirt package in R software (Chalmers, 2012). Rasch analysis of the baseline data resulted in dropping one item ("Do you allow this child to play-fight, testing who is strongest?") due to local dependence. Theta standardized scores from the Rasch analysis of the final 30-item TRiPS total scale ranged from -3.372 to 1.975, with a mean of 0.000 (SD 0.974). A higher standardized score indicates higher tolerance of risky outdoor play.
Time Frame: Baseline, 1-week-post-intervention, 3-month-post-intervention
Population: Included was 451 mothers with baseline demographic data; and, 351 mothers with baseline outcome data (TRiPS) at baseline, 333 mothers at 1-week-post-intervention, and 312 mothers at 3-month-post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Position Statement on Active Outdoor Play: Position Statement Active Outdoor Play: The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety (ParticipACTION, 2015; Tremblay et al., 2015).
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool | RR In-Person Workshop
Number analyzed (Participants) | 148 | 150 | 153
score on a scale
  Baseline outcome: number analyzed (Participants) | 145 | 121 | 85
  Baseline outcome | 0.05 (1.03) | -0.14 (0.97) | 0.18 (0.87)
  1-week-post-intervention outcome: number analyzed (Participants) | 135 | 113 | 85
  1-week-post-intervention outcome | -0.09 (1.03) | -0.06 (1.05) | 0.22 (0.80)
  3-month-post-intervention outcome: number analyzed (Participants) | 123 | 105 | 84
  3-month-post-intervention outcome | -0.03 (0.92) | -0.09 (0.93) | 0.15 (0.80)

2. Secondary Outcome: Self-reported Behaviour Change
Description: The secondary outcome measure was self-reported behavior change, measured by participants' self-reported progress on attaining the goal they set for themselves within the risk reframing intervention. At each follow-up, participants were reminded of their goal (by asking "at the beginning of the study, you set a goal for yourself regarding something you wanted to change to give your child more opportunities for risky play. Have you made progress toward this goal?") and asked "Did you accomplish your goal?" with "Yes" and "No" response options. For the purpose of our analyses the category of "Yes" is an indication of behaviour change while the category of "No" is an indication of no behaviour change.
Time Frame: 1-week-post-intervention, 3-month-post-intervention
Population: Included was 333 mothers with complete secondary outcome data (Goal) at 1-week post-intervention - which represents the first time we collected these data; and 312 mothers at 3-month-post intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool | RR In-Person Workshop
Number analyzed (Participants) | 135 | 113 | 85
Participants
  1-week-post-intervention participants who responded: Yes | 76 | 81 | 47
  1-week-post-intervention participants who responded: No | 59 | 32 | 38
  3-month-post-intervention participants who responded: number analyzed (Participants) | 123 | 105 | 84
  3-month-post-intervention participants who responded: Yes | 99 | 90 | 62
  3-month-post-intervention participants who responded: No | 24 | 15 | 22

ADVERSE EVENTS:
Description: Adverse events were not monitored/assessed because this RCT was not clinical-based. It was to test the efficacy of a web-based intervention to change participants' perception of risk in children's outdoor play.
Arm/Group | Risk Reframing (RR) Digital Tool | RR In-Person Workshop | Position Statement on Active Outdoor Play
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Given the nature of the interventions, it was not possible to blind participants to their allocation, thus potentially introducing sources of bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT03374683/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03374683/ICF_001.pdf